CLINICAL TRIAL: NCT05115617
Title: Pregnant and Lactating Individuals & Newborns COVID-19 Vaccination (PLAN-V): Prospective Cohort Study
Brief Title: Pregnant and Lactating Individuals & Newborns COVID-19 Vaccination Prospective Cohort Study
Acronym: PLAN-V
Status: Recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital of Eastern Ontario Research Institute (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Darine El-Chaâr, Principal Investigator, Ottawa Hospital Research Institute
Other Study IDs: CTO 3612
Record Dates: First submitted 2021-09-28; First posted 2021-11-10 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV2 Infection; Covid19; Vaccine Reaction; Pregnancy Related; Immunogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Should residual samples (i.e. maternal serum, umbilical cord serum, breast milk, placental tissue [frozen and fixed]) remain after the purposes of the primary outcomes, samples will be retained for up to 25 years for future, related REB approved studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant individuals: Pregnant individuals who have previously received one-dose of COVID-19 vaccine, or who are planning to receive a COVID-19 vaccine in pregnancy.

SUMMARY:
The PLAN-V Study is an Ontario-based prospective, longitudinal study that will consist of extensive biosampling and detailed data collection from pregnant women/individuals, who have received the COVID-19 vaccine during their pregnancy, and their infants across the antenatal, delivery and postpartum periods.

DETAILED DESCRIPTION:
There is a pressing need for research to answer critical questions about the role of maternal vaccination for protection of the mother-infant dyad, to inform public health recommendations and to support evidence-based decision-making by Canadian families and their care providers.

The investigators' goal is to generate rapid, reliable evidence specific to the immunogenicity and safety of COVID-19 vaccines in the pregnant population. The specific PLAN-V Study objectives are:

1. To evaluate immunogenicity of COVID-19 vaccines in pregnant women/individuals and the fetal/newborn immune response to maternal vaccination.
2. To evaluate safety of COVID-19 vaccination in pregnant women/individuals based on obstetrical, fetal and newborn health outcomes.
3. To compare immune responses to COVID-19 vaccination and natural COVID-19 disease among pregnant women/individuals and their infants exposed in utero
4. To compare the immune responses to COVID-19 vaccination between pregnant and non-pregnant women/individuals.

PLAN-V is an Ontario-based prospective, longitudinal study that will consist of extensive biosampling and detailed data collection from pregnant women/individuals and their infants across the prenatal, delivery and postpartum periods. With this approach, detailed participant profiles will be generated that will enable us to explore vaccine reactogenicity; vaccine-associated adverse events; frequency of obstetrical and fetal/newborn outcomes; and measures of infant health and well-being. The study will build on existing resources and expertise available through the COVID-19 Ontario Pregnancy Event (COPE) Network to establish a prospective, longitudinal cohort study of pregnant women/individuals, and their infants.

The PLAN-V Study will consist of pregnant women/individuals who are planning to receive a COVID-19 vaccine(s) at any stage in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women/Individuals ≥ 16 years of age who are ≥7 0/7 weeks' gestation on the day of enrollment
* Capacity to provide informed consent and to comprehend and comply with the study requirements
* Planning to deliver at a participating site hospital
* Planning to receive or have previously received one-dose of a Health Canada approved COVID-19 vaccine (any product, any number of doses) during the current pregnancy

Exclusion Criteria:

* Cases with known major fetal concerns
* Women/Individuals who are fully vaccinated against COVID-19
* Women/Individuals who are pregnant due to surrogacy, or planning to give their child up for adoption
* Women/Individuals with a non-viable pregnancy (e.g., ectopic)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The PLAN-V Study will consist of pregnant women/individuals who are planning to receive a COVID-19 vaccine(s) at any stage in pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Antibody titres in biological samples | 1-month post COVID-19 vaccine
  Immunogenicity of COVID-19 Vaccines: Seroconversion rates in vaccinated mothers, SARS-CoV-2 antibody titres and their persistence in mothers after vaccination in pregnancy, transfer of antibodies to breastmilk/chestmilk, transfer and persistence of SARS-CoV-2 antibodies to the neonate/infant over the study period.
Antibody titres in biological samples | 3-month, and 6-month post COVID-19 vaccine
  Immunogenicity of COVID-19 Vaccines: Seroconversion rates in vaccinated mothers, SARS-CoV-2 antibody titres and their persistence in mothers after vaccination in pregnancy, transfer of antibodies to breastmilk/chestmilk, transfer and persistence of SARS-CoV-2 antibodies to the neonate/infant over the study period.
Antibody titres in biological samples | 6-month post COVID-19 vaccine
  Immunogenicity of COVID-19 Vaccines: Seroconversion rates in vaccinated mothers, SARS-CoV-2 antibody titres and their persistence in mothers after vaccination in pregnancy, transfer of antibodies to breastmilk/chestmilk, transfer and persistence of SARS-CoV-2 antibodies to the neonate/infant over the study period.
Antibody titres in biological samples | At delivery
  Immunogenicity of COVID-19 Vaccines: Seroconversion rates in vaccinated mothers, SARS-CoV-2 antibody titres and their persistence in mothers after vaccination in pregnancy, transfer of antibodies to breastmilk/chestmilk, transfer and persistence of SARS-CoV-2 antibodies to the neonate/infant over the study period.
Antibody titres in biological samples of participants who received COVID-19 vaccine and who had natural COVID-19 disease. | 6-months post-COVID-19 vaccine
  Comparing immune responses to COVID-19 vaccination in pregnant and non-pregnant women/individuals
Antibody titres in biological samples of participants who received COVID-19 vaccine and who had natural COVID-19 disease. | 3-month post-COVID-19 vaccine
  Comparing immune responses to COVID-19 vaccination in pregnant and non-pregnant women/individuals
Antibody titres in biological samples of participants who received COVID-19 vaccine and who had natural COVID-19 disease. | 1-month post-COVID-19 vaccine
  Comparing immune responses to COVID-19 vaccination in pregnant and non-pregnant women/individuals
Antibody titres in biological samples of pregnant and non-pregnant populations | During delivery admission
  Comparing infection-acquired and vaccine-acquired immunity against COVID-19 in mothers and newborns

SECONDARY OUTCOMES:
Maternal death | through study completion, an average of 9 months
  Maternal death during delivery admission
Maternal - Non-delivery hospitalization | through study completion, an average of 9 months)
  Any hospitalization not associated with the delivery of infant.
Any infection | through study completion, an average of 9 months
  Maternal diagnosis of any infection during pregnancy
Pre-term labour | through study completion, an average of 9 months
  The onset of labour prior to 37 weeks gestation
Hypertensive disorders of pregnancy | through study completion, an average of 9 months
  The diagnosis of a hypertensive disorder of pregnancy
Placental abruption | through study completion, an average of 9 months
  The diagnosis of placental abruption during pregnancy
Postpartum hemorrhage | Post-delivery, during the delivery admission
  The diagnosis of postpartum hemorrhage
Preterm birth | through study completion, an average of 9 months
  Infant born prior to 37 weeks gestation
Fetal loss or stillbirth | through study completion, an average of 9 months
  Fetal loss or stillbirth throughout the pregnancy
Small for gestational age | During the pregnancy, through study completion, an average of 9 months
  <10th percentile for gestational age and sex- specific birth weight
Term low birthweight | At delivery
  <2500g
Low 5 min Apgar Score | At delivery
  Score <5 at 5 minutes
Low cord blood pH | At delivery
  cord blood pH<7.0
admission to neonatal ICU for >12 hours | During delivery admission
  Infant admission to the neonatal ICU for >12 hours
composite neonatal adverse outcome indicator [NAOI] | At delivery
  A composite indicator which includes various neonatal adverse outcomes
Frequency of infection | Postpartum, through study completion, an average of 9 months
  Number of infections, including but not limited to: influenza, pneumonia, sepsis, acute respiratory infections, gastrointestinal
Re-hospitalization rates | Postpartum, through study completion, an average of 9 months
  Number of re-hospitalizations and emergency visits
Composite indicator for complex chronic conditions | Postpartum, through study completion, an average of 9 months
  Composite indicator includes: neurologic and neuromuscular; cardiovascular; respiratory; renal and urologic; gastrointestinal; hematologic or immunologic; metabolic; other congenital or genetic defect; and malignancy
Infant death | Postpartum, through study completion, an average of 9 months
  Infant death

CONTACTS AND LOCATIONS:
Overall Officials: Darine El-Chaâr, MD, MSc, Principal Investigator — The Ottawa Hospital
Locations (7):
- Canada (7):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - The Ottawa Hospital - General, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD that underlie the results reported in this article, after deidentification, will be made available to other researchers upon request.

DOCUMENTS (1):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT05115617/Prot_000.pdf